CLINICAL TRIAL: NCT07115433
Title: Effectiveness of a School-Based Oral Health Promotion Program on Oral Health Practices, Behaviour, Self-Efficacy, and Clinical Outcomes Among Primary School Children: A Randomized Controlled Trial
Brief Title: Effectiveness of School-based Oral Health Intervention for Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Arshed Muhammad, PhD, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: BMU-BDC
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Oral; Health

STUDY DESIGN:
Intervention Model Description: It is two arm randomized control trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and outcome assessors will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group will be given no intervention other than they will receive routinely
- Intervention group (Experimental): Arm Description: The oral health promotion intervention will be implemented through weekly interactive sessions lasting 30-40 minutes over a period of six months. These sessions, conducted by trained dental educators and teachers, will use animations, storytelling, demonstrations, and role-plays to teach proper toothbrushing, the importance of fluoride toothpaste, healthy eating habits, and the need for regular dental visits. Children will participate in supervised toothbrushing once a week, supported by peer ambassadors who reinforce daily practices. Educational leaflets and videos will engage parents, while posters in classrooms serve as reminders. Follow-up assessments, including questionnaires and clinical indices, will be conducted at six months.
  Interventions: Behavioral: School-Based Oral Health Promotion Program

INTERVENTIONS:
Behavioral: School-Based Oral Health Promotion Program — Arm Description: The oral health promotion intervention will be implemented through weekly interactive sessions lasting 30-40 minutes over a period of six months. These sessions, conducted by trained dental educators and teachers, will use animations, storytelling, demonstrations, and role-plays to teach proper toothbrushing, the importance of fluoride toothpaste, healthy eating habits, and the need for regular dental visits. Children will participate in supervised toothbrushing once a week, supported by peer ambassadors who reinforce daily practices. Educational leaflets and videos will engage parents, while posters in classrooms serve as reminders. Follow-up assessments, including questionnaires and clinical indices, will be conducted at six months.
  Arms: Intervention group

SUMMARY:
Schools provide an ideal setting for early interventions. Evidence suggests that educational programs incorporating behavioural change theories can improve oral hygiene practices and clinical outcomes.

A School-Based Oral Health Promotion Program on Oral Health Practices, Behaviour, Self-Efficacy, and Clinical Outcomes Among Primary School Children for six months, while the control group will receive no intervention, only routine care.

DETAILED DESCRIPTION:
Poor oral health in children leads to pain, absenteeism, and impaired quality of life. Schools provide an ideal setting for early interventions. Evidence suggests that educational programs incorporating behavioural change theories can improve oral hygiene practices and clinical outcomes.

A School-Based Oral Health Promotion Program on Oral Health Practices, Behaviour, Self-Efficacy, and Clinical Outcomes Among Primary School. The oral health promotion intervention will be implemented through weekly interactive sessions lasting 30-40 minutes over six months. These sessions, conducted by trained dental educators and teachers, will use animations, storytelling, demonstrations, and role-plays to teach proper toothbrushing, the importance of fluoride toothpaste, healthy eating habits, and the need for regular dental visits. Children will participate in supervised toothbrushing once a week, supported by peer ambassadors who reinforce daily practices. Educational leaflets and videos will engage parents, while posters in classrooms serve as reminders. Follow-up assessments, including questionnaires and clinical indices, will be conducted at six months, while the control group will receive no intervention, only routine care.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-8 years enrolled in selected schools
* Written informed consent from parents/guardians and assent from children

Exclusion Criteria:

* Children with systemic conditions affecting oral health
* Those currently in other oral health interventions

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Plaque score | 6 months
  Plaque score index: 0: No plaque.
  1. Separate flecks of plaque at the gum line.
  2. A thin band of plaque along the gum line.
  3. A band of plaque wider than 1mm but covering less than one-third of the tooth.
  4. Plaque covering one-third to two-thirds of the tooth.
  5. Plaque covering more than two-thirds of the tooth. Higher scores indicate more plaque and poorer oral hygiene.
Oral Hygiene | 6-months
  Oral Hygiene will be assessed by the presence of debris (plaque) and calculus (tartar) on selected tooth surfaces, measured by the Simplified Oral Hygiene Index (OHI-S)
  Individual Debris Index (DI-S) and Calculus Index (CI-S):
  Each of the six surfaces is scored individually for both debris and calculus using a 0-3 scale:
  0: No debris or calculus is present.
  1. Debris or calculus covers less than one-third of the surface.
  2. Debris or calculus covers between one-third and two-thirds of the surface.
  3. Debris or calculus covers more than two-thirds of the surface. Good: 0.0 - 1.2 Fair: 1.3 - 3.0 Poor: 3.1 - 6.0
Gingival score | 6 months
  Gingival score assessed by the gingival score index:
  0: Normal gingiva, no inflammation.
  1. Mild inflammation - slight color change and edema (swelling), no bleeding on probing.
  2. Moderate inflammation - redness, edema, glazing, and bleeding on probing.
  3. Severe inflammation - marked redness, edema, ulceration, and tendency towards spontaneous bleeding. The index typically uses a scale of 0 to 3, with 0 representing normal gingiva and higher scores indicating increasing severity of inflammation

SECONDARY OUTCOMES:
oral health practices | 6 months
  Oral health practices by using the WHO Child Oral Health Questionnaire: o assess children's oral health practices through a structured set of questions. These questionnaires typically cover knowledge, attitude, and practices related to oral hygiene, including frequency of brushing, use of fluoride toothpaste, and dental visits. The score is used to evaluate the overall oral health practices of the child, often categorized as good, fair, or poor.
Oral Health Impact Profile. | 6 months
  Oral Health Impact Profile. The Oral Health Impact Profile (OHIP) is a questionnaire used to assess how oral health problems affect a person's daily life and well-being. The OHIP-14, a shorter version, is commonly used and focuses on 14 specific questions related to oral health impacts 0 = Never
  1. = Hardly ever
  2. = Occasionally
  3. = Fairly often
  4. = Very often Greater score shows better impact andvice versa

CONTACTS AND LOCATIONS:
Locations (3):
- Pakistan (3):
  - Saleem ullah fahmi school baqai Medical complex gharo, Karachi, Sindh
  - Saleem ullah fahmi memorial school unit 1, Karachi
  - Saleem ullah fahmi school Khuda ki basti, Karachi

IPD SHARING:
Plan to Share IPD: No
Only the study protocol, statistical plan, and results will be shared in publications in peer-reviewed journals

REFERENCES:
- [Background] nsari Moghaddam S, Shahrzad S, Kermansaravi F. Effect of teach-back method on oral health indicators, self-efficacy, and self-care behaviors of high school students in Zahedan during 2019. J Mashhad Dent School. 2020;44(2):99-113.
- [Background] Hashemi ZS, Khorsandi M, Shamsi M, Moradzadeh R. Effect combined learning on oral health self-efficacy and self-care behaviors of students: a randomized controlled trial. BMC Oral Health. 2021 Jul 13;21(1):342. doi: 10.1186/s12903-021-01693-y. PMID 34256752
- [Background] Sanaeinasab H, Saffari M, Taghavi H, Karimi Zarchi A, Rahmati F, Al Zaben F, Koenig HG. An educational intervention using the health belief model for improvement of oral health behavior in grade-schoolers: a randomized controlled trial. BMC Oral Health. 2022 Mar 27;22(1):94. doi: 10.1186/s12903-022-02132-2. PMID 35346148
- [Background] Hernandez-Vasquez A, Azanedo D. The urgency of ensuring equitable and improved access to oral health care during the Coronavirus Disease 2019 pandemic: The case of Peru. J Res Health Sci. 2021 Aug 28;21(3):e00528. doi: 10.34172/jrhs.2021.60. PMID 34698662